CLINICAL TRIAL: NCT02707471
Title: Improving Well-Being for Breast Cancer Patients Taking Adjuvant Endocrine Therapy
Brief Title: Improving Well-Being for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00068595
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Self-management Intervention (SM-AET); General Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SM-AET (Experimental): a self-management intervention for enhancing skills to improve adherence and reduce symptom interference (SM-AET) (active intervention group)
  Interventions: Behavioral: SM-AET
- general health education Intervention (Other): general health education Intervention (control group)
  Interventions: Behavioral: general health education

INTERVENTIONS:
Behavioral: SM-AET — self-management for improving adherence and reducing symptom interference (SM-AET)
  Arms: SM-AET
Behavioral: general health education — general health education intervention that focuses on improving overall health.
  Arms: general health education Intervention

SUMMARY:
Adjuvant endocrine therapy (AET) is a crucial component of treatment used to prevent recurrence and reduce breast cancer-related mortality for breast cancer patients with hormone receptor positive disease. Studies report low rates of adherence to AET (38% to 86%) and in our preliminary work, 65% of breast cancer patients taking AET reported one or more non-adherent medication taking behaviors (e.g., skipped dose, forgot, adjusted dose) in the past month. Symptoms (e.g., arthralgia, vasomotor symptoms) associated with AET are strongly related to non-adherence and early discontinuation of treatment. Poor adherence to AET due to symptoms may compromise the effectiveness of AET. Prior to conducting a clinical trial, we will conduct user testing of the self-management intervention protocol with 20 women. In the proposed randomized clinical trial, 400 women who are taking AET for breast cancer will be randomly assigned to one of two conditions: 1) a self-management intervention for improving adherence and symptom management, or 2) a general health education control condition. The self-management intervention integrates three key theory-based strategies for improving adherence to AET: coping skills training for managing symptoms (e.g., arthralgia, vasomotor symptoms), behavioral strategies for improving medication adherence, and symptom and medication education. The intervention addresses the specific symptoms a woman is experiencing and is designed to meet the needs of women who are at high risk for non-adherence to AET (e.g., low socioeconomic status, low literacy). The self-management intervention is administered by a nurse via the telephone, and combines the use of phone calls and tailored interactive voice messaging based on information exchanged during phone sessions and real-time adherence data obtained from smart medication bottles. Women randomly assigned to the control condition will receive a general health education intervention that is delivered by a nurse via the telephone. This study will take place in the Duke Cancer Institute breast clinic and in community hospitals that are members of the Duke Cancer Network, which will allow access to women receiving care outside the medical center setting and increase generalizability of findings to a variety of settings. Adherence to AET will be assessed over the 18 month period following study enrollment using wireless smart medication bottles that provide real-time adherence data and pill counts completed by study staff during in-person study assessments. Patient-reported outcome measures assessing symptoms, perceived necessity of AET, concerns about AET, and self-efficacy will be obtained at baseline and 3, 6, 12, and 18 months. To increase the likelihood of later implementation of the self-management intervention, the cost effectiveness of the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Stage I to III breast cancer
* hormone receptor positive tumor defined as any positivity of estrogen or progesterone receptor
* completed local definitive treatment (i.e., surgery, chemotherapy, radiation),
* within 12 months of beginning AET
* at least 18 months of AET recommended

Exclusion Criteria:

* <21 years of age,
* severe cognitive or hearing impairment that is documented in the medical record
* unable to provide meaningful consent (e.g., severe cognitive impairment).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Percent daily adherence assessed over 18 months | 18 month
  The SM-AET protocol includes eight sessions and two maintenance calls administered by a nurse via the phone. The intervention also includes interactive voice messaging that is tailored based on participants' medication taking behavior. Adherence to AET will be assessed using smart pill bottles (i.e., bottle opening and percent of pills remaining).

SECONDARY OUTCOMES:
Change in medication taking behaviors | Baseline, 3 months, 6 months, 12 months, 18 months
  A revised 16-item measure based on the Medication Adherence Rating Scale and our prior studies is used to assess self-reported adherence. Items were revised to refer specifically to participants' AET medication, assess medication-taking behaviors related to adherence (e.g., forgetting), and capture intentional and unintentional nonadherence over the past month.
Change in Menopausal Symptoms and Symptom Interference | Baseline, 3 months, 6 months, 12 months, 18 months
  The 32-item Menopause Specific Quality of Life Questionnaire (MENQOL) assesses the degree of symptom interference in the past week related to four domains: physical symptoms, vasomotor symptoms, psychosocial symptoms, and sexual symptoms.
Change in Pain and Joint Stiffness/Aching and Symptom Interference | Baseline, 3 months, 6 months, 12 months, 18 months
  The Brief Pain Inventory - Short form (BPI-SF) is used to assess pain interference in the past week across 9 areas (e.g., general activity, mood, sleep, enjoyment of life). Five items adapted from the Arthritis Impact Measurement Scale-II (AIMS-II; e.g., How would you describe the joint aching that you usually had?; How often did joint aching make it difficult to sleep?) and four items modified from the BPI-SF pain severity scale (e.g., Please rate stiffness in your joints by selecting the one number that best describes your stiffness at its worst in the past week) are used to measure aching and joint stiffness.
Change in Sleep Problems | Baseline, 3 months, 6 months, 12 months, 18 months
  The 7-item Insomnia Severity Index (ISI) is a measure of participants' perceived severity of sleep difficulties and the interference of these difficulties with emotional distress, daily functioning, and quality of life in the last two weeks.
Change in Fatigue | Baseline, 3 months, 6 months, 12 months, 18 months
  The 8-item Patient Reported Outcomes Information System Fatigue Scale (PROMIS Fatigue) assesses fatigue over the past seven days.
Change in psychological distress | Baseline, 3 months, 6 months, 12 months, 18 months
  The eight-item Patient Reported Outcomes Information System Depression Scale (PROMIS Depression) assesses depressive symptoms. The eight-item Patient Reported Outcomes Information System Anxiety Scale (PROMIS Anxiety) is used to assess symptoms of anxiety.
Change in Physical Functioning and Symptom Interference: 6-minute walk test | Baseline, 3 months, 6 months, 12 months, 18 months
  The 6-minute walk test assesses women's abilities to exert effort in activity and the degree of pain experienced during activity. Women are asked to walk along an indoor hallway for 6-minutes with the goal being to walk as far as possible within the allotted time. Total distance in feet walked during the allotted time is recorded.
Change in Physical Functioning and Symptom Interference: Get Up and Go test | Baseline, 3 months, 6 months, 12 months, 18 months
  In the timed get up and go test participants are asked to stand up from a chair, walk 10 feet, turn, walk back to the chair, and sit down. Total time to complete the task is recorded in seconds.
Change in Physical Functioning and Symptom Interference: Grip strength | Baseline, 3 months, 6 months, 12 months, 18 months
  Grip strength is assessed using a latex free JAMAR hydraulic hand dynamometer. The participant sits with her forearm in a neutral position, and wrist between 0° and 30° dorsiflexion and between 0° and 15° ulnar deviation. She then squeezes the handle of the dynamometer as hard as she can. Data is recorded in pounds. Three trials are conducted with each hand.
Change in perceived barriers to taking AET medication | Baseline, 3 months, 6 months, 12 months, 18 months
  Eleven items assess barriers to taking medication over the past month. Specifically, women rate how often certain situations (e.g., forgetfulness, problematic side effects, being out of routine) make it difficult for them to take their medications every day.
Change in treatment interference | Baseline, 3 months, 6 months, 12 months, 18 months
  Five items from the Treatment Burden Questionnaire assess how often, time spent, frequency, or inconveniences associated with recommended health care present a problem for the participant.
Change in beliefs about medication | Baseline, 3 months, 6 months, 12 months, 18 months
  The 10-item Beliefs about Medicines Questionnaire (BMQ) assesses perceived necessity and concerns about AET (e.g., my health depends on my medicine, my medicine protects me from becoming ill).
Change in self-efficacy for managing symptoms and taking AET | Baseline, 3 months, 6 months, 12 months, 18 months
  An 8-item scale will measure self-efficacy for managing symptoms. Participants are asked to rate how confident they are that they can manage common symptoms (e.g., aches and plain, sexual side effects and hot flashes/sweating) related to AET. The 13-item Self-Efficacy for Appropriate Medication Use Scale assesses self-efficacy for taking medications across various situations (e.g., when no one reminds you to take the medicine, when you have a busy day planned, when you are away from home).
Estimate of cost-effectiveness of the CST-AET intervention | Baseline, 3 months, 6 months, 12 months, 18 months
  The 5-level EuroQol-5 Dimensions (EQ-5D-5L) health questionnaire assesses current health status across five domains that map to a 0 (dead) to 1 (perfect health) scale representing the relative utility (or desirability) of health-related quality of life. These utility weights are used to derive quality-adjusted life years (QALYs).

OTHER OUTCOMES:
Treatment Credibility and Satisfaction | 3 months, 6 months
  The Treatment Crediblity Questionnaire is a 5-item measure of the degree to which participants perceive a treatment as credible and expect positive outcomes (e.g., how helpful does the therapist seem to you?; how confident are you that this treatment will help you manage your symptoms and health concerns?). The Satisfaction with Therapy and Therapist Scale is a 13-item measure that has been modified to obtain participants' satisfaction with the intervention and the nurse delivering the intervention sessions. Items assess satisfaction with and global improvement (i.e., how much did the intervention help with your symptoms and health concerns) after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Shelby RA, Dorfman CS, Bosworth HB, Keefe F, Sutton L, Owen L, Corsino L, Erkanli A, Reed SD, Arthur SS, Somers T, Barrett N, Huettel S, Gonzalez JM, Kimmick G. Testing a behavioral intervention to improve adherence to adjuvant endocrine therapy (AET). Contemp Clin Trials. 2019 Jan;76:120-131. doi: 10.1016/j.cct.2018.11.010. Epub 2018 Nov 22. PMID 30472215

DOCUMENTS (1):
  • Informed Consent Form (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02707471/ICF_000.pdf